CLINICAL TRIAL: NCT05950984
Title: An Investigation Into How Medical Device Obtained Variables Influence the Pharmacokinetic Profile of Vancomycin: a Paediatric and Adult Critical Care Feasibility Assessment at a London Tertiary-care Hospital
Brief Title: Medical Device (MD) Derived Pharmacokinetic (PK) Parameters for Vancomycin (MD-PK)
Acronym: MD-PK
Status: Completed | Type: Observational
Sponsor: St George's, University of London (Other)
Collaborators: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 2022.0286
Record Dates: First submitted 2023-05-29; First posted 2023-07-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2024-01

CONDITIONS: Infection, Bacterial; Antibiotic Side Effect; Antibiotic Resistant Infection; Sepsis; Septic Shock; Bacteremia; Critical Illness; Adult Children
Keywords: Vancomycin; Pharmacokinetics; Accuracy; Medical Device; Digital; Data; Protein Binding; Critical Illness; Drug Infusion Pump; Electronic Prescribing and Administration System; Point of Care; Therapeutic Drug Monitoring
MeSH Terms: conditions — Bacterial Infections; Sepsis; Shock, Septic; Bacteremia; Critical Illness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Critically Ill Adults and Children: Adults and children from 1-day old admitted to a critical care unit.
  Interventions: Other: Drug Infusion Pump Monitoring

INTERVENTIONS:
Other: Drug Infusion Pump Monitoring — Intravenous vancomycin administration accuracy will be determined by comparing data obtained from drug infusion pumps with manually input administration times from the electronic Prescribing and Medicines Administration (ePMA) system.

SUMMARY:
Getting the right dose of antibiotic promptly is an important part of treating infections. Unfortunately, when an infection is severe (sepsis) the body changes how it processes antibiotics. Consequently, some people with severe infection retain antibiotics for too long (risking adverse effects), whilst others excrete antibiotics too quickly (risking under-treatment).

Mathematical models can help researchers understand drug handling variability (known as pharmacokinetics) between people. These models require very accurate information about drug administration and drug blood concentration timings. Researchers usually rely on someone recording these timings, but recording errors can make models inaccurate.

We would like to understand if using data from routinely used electronic drug infusion devices (recording the exact time of administration) can improve the accuracy of pharmacokinetic models. We intend to investigate this with an antibiotic (vancomycin) that clinicians already routinely monitor blood concentrations for. Adults and children treated at St George's Hospital intensive care units will be invited to participate in the study which will last for 28-days within a 14-month period. Participants will donate a small amount of extra blood and provide researchers access to their clinical data. Blood will be taken at special times during vancomycin treatment from lines placed as part of standard treatment, minimising any pain or distress. There will be no other changes to patient's treatment.

In the future, data from this study might help change the way we dose antibiotics. The National Institute for Health and Care Research and Pharmacy Research UK are supporting the study with funding.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to either adult or paediatric intensive care unit (ICU) and receiving intravenous vancomycin (continuous or intermittent infusion only), to prevent or treat a clinical infection
* Informed consent form signed by participant/parent/legal guardian/legal representative (as determined by age group/capacity, consent may be retrospective) or signed informed personal/nominated consultee declaration
* Age from 1-day since birth

Exclusion Criteria:

* Previous enrolment into this study
* Treating clinician feels participant unlikely to survive beyond 48-hours from enrolment or treatment has been withdrawn for reasons of palliation
* Absence of in-dwelling vascular access from which samples may be drawn or removal of in-dwelling access prior to retrieval of a 3rd blood sample (for assay of vancomycin concentration)
* Non-continuous renal replacement (i.e. intermittent haemodialysis/ peritoneal dialysis)
* Hypersensitivity or allergies to vancomycin, its excipients, or the infusion fluid
* Treatment outside an ICU area

In paediatrics:

* Required blood sampling exceeds 3% of total blood volume in a four-week period or 1% at any single time (European Medicines Agency, 2009)
* Where there is disagreement between child consent/assent and parental/ legal guardian consent/assent

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults and children admitted to an intensive care unit and administered intravenous vancomycin for prevention/treatment of an infection
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2024-08-28 (Actual)

PRIMARY OUTCOMES:
Objective Function Value | Within collection of 15 vancomycin serum concentrations or 28 days from first study recorded administration of vancomycin
  Pharmacokinetic model fit determined quantitively by Objective Function Value (2.log likelihood) using vancomycin administration time data recorded by patient's bedside drug infusion devices compared to manually recorded data

SECONDARY OUTCOMES:
Participant Vancomycin Volume of Distribution | Within collection of 15 vancomycin serum concentrations or 28 days from first study recorded administration of vancomycin
  Calculation of participant's vancomycin volume of distribution (litres) using non-linear mixed effects modelling methods from obtained non-protein bound and total vancomycin concentrations and patient's drug infusion device obtained administration time data
Participant Vancomycin Clearance | Within collection of 15 vancomycin serum concentrations or 28 days from first study recorded administration of vancomycin
  Calculation of participant vancomycin clearance (litres/hour) using non-linear mixed effects modelling methods using obtained non-protein bound and total vancomycin concentrations and participant's drug infusion device derived administration time data
Participant 24-hour Area Under the Vancomycin Concentration Time Curve (AUC) | Within collection of 15 vancomycin serum concentrations or 28 days from first study recorded administration of vancomycin
  Calculation of participant's AUC (milligrams.hour/litre) using obtained non-protein bound and total vancomycin concentrations and participant's drug infusion device derived administration time data
Participant 24-hour AUC:MIC Ratio | Within collection of 15 vancomycin serum concentrations or 28 days from first study recorded administration of vancomycin
  Calculation of the area under the 24-hour non-protein bound and total vancomycin concentration AUC/bacterial minimum inhibitory concentration (MIC) ratio using an empiric MIC of 1mg/L or MIC of obtained isolates (if available) using trapezial rule or vancomycin dose and calculated clearance

OTHER OUTCOMES:
Association Between Participant's Mean 24-hour AUC:MIC and Microbiological Cure | Within collection of 15 vancomycin serum concentrations or 28 days from first study recorded administration of vancomycin
  Microbiological cure defined as eradicated baseline microorganisms and no new microorganisms are identified via bacterial cultures (if available), plus, the patient has received allocated treatment for at least 2-days with no modification or a failure
Association Between Participant's Mean 24-hour AUC:MIC and Length of Intensive Care (ICU) Unit Stay | Within collection of 15 vancomycin serum concentrations or 28 days from first study recorded administration of vancomycin
  ICU stay quantified by days since admission, categories include: <2 days, < 7 days, <14 days, >14 days
Association Between Participant's Mean 24-hour AUC:MIC and Infection Related Mortality | Within collection of 15 vancomycin serum concentrations or 28 days from first study recorded administration of vancomycin
  Cause of mortality will be derived from participant's medical notes
Association Between Participant's Mean 24-hour AUC:MIC and Infection related ICU Re-admission | Within collection of 15 vancomycin serum concentrations or 28 days from first study recorded administration of vancomycin
  Cause of re-admission will be derived from participant's medical notes
Association Between Participant's Mean 24-hour AUC:MIC and Vancomycin Associated Acute Kidney Injury (AKI) | Within collection of 15 vancomycin serum concentrations or 28 days from first study recorded administration of vancomycin
  AKI defined by Kidney Disease: Improving Global Outcomes (KDIGO) Criteria
Association Between Participant's Mean 24-hour AUC:MIC and Adult National Early Warning Score (NEWS2) or Paediatric Early Warning Score (PEWS3) | Within collection of 15 vancomycin serum concentrations or 28 days from first study recorded administration of vancomycin
  Warning scores calculated on day of (and closest to) first dose of study recorded vancomycin treatment course, between 2-3 days since vancomycin course initiation and at end of vancomycin course or 28 days from first study recorded administration of vancomycin

CONTACTS AND LOCATIONS:
Locations (1):
- St Georges University Hospitals NHS Foundation Trust, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Fully anonymised collected patient data may be shared if consent provided with select research collaborators

REFERENCES:
- [Background] Oakley R, Bakrania P, Yau T, Standing J, Lonsdale D. Variable adherence to and effectiveness of a vancomycin continuous infusion protocol within ICUs at a London tertiary-care hospital: a single-centre retrospective service evaluation 2022;4:dlac004.036. https://doi.org/10.1093/jacamr/dlac004.036
- [Background] Correction to: Improving adherence to and effectiveness of an adult critical care vancomycin continuous infusion protocol: a pilot quality improvement and administration data accuracy project. JAC Antimicrob Resist. 2023 Jun 8;5(3):dlad075. doi: 10.1093/jacamr/dlad075. eCollection 2023 Jun. PMID 37305849